CLINICAL TRIAL: NCT04211922
Title: A Phase II, Multicenter, Single-arm Study to Evaluate Safety and Efficacy of Alkotinib Capsule in Patients With ALK-positive Non-small Cell Lung Cancer Previously Treated With Crizotinib
Brief Title: Alkotinib Capsule in Patients With ALK-positive Non-small Cell Lung Cancer Previously Treated With Crizotinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor R&D Strategy Adjustment
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGALK002
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: ALK-positive Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alkotinib 400mg QD (Experimental): 400mg orally once daily. Take Alkotinib at least 1 hour before or at least 2 hours after a meal.
  Interventions: Drug: Alkotinib Capsules

INTERVENTIONS:
Drug: Alkotinib Capsules — Alkotinib 400mg QD
  Other Names: ZG0418

SUMMARY:
The main purpose of the study is to evaluate safety and efficacy of Alkotinib capsule in patients with ALK-positive non-small cell lung cancer previously treated with crizotinib.While exploring the relationship between biomarkers and drug efficacy and safety.

DETAILED DESCRIPTION:
The drug being tested in this study is called alkotinib. Alkotinib has been demonstrated to benefit people with ALK+ NSCLC.

The study is a non-control study.

The study will enroll approximately 104 participants. All participants will take alkotinib 300mg throughout the study.

This multi-center trial will be conducted in China. The overall time to participate in this study is 3 years. Participants will make multiple visits to the site, and 28 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of positive ALK.
* Patients must have demonstrated progression during or after crizotinib treatment.
* Age 18 years or older at the time of informed consent.
* Eastern cooperative oncology group performance status (ECOG PS) of 0-2
* At least one measurable lesion by response evaluation criteria in solid tumors (RECIST) version 1.1 (v1.1).
* Willingness and ability to comply with the trial and follow-up procedures.

Exclusion Criteria:

* chemotherapy, radiation therapy, immunotherapy within 4 weeks.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of study medications.
* Uncontrolled mass of pleural effusion, pericardial effusion, and peritoneal effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on independent radiology review | 24 months
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) as assessed by independent radiology review and investigator | 36 months
  PFS, defined as time from first dose of Alkotinib to progression or death due to any cause.
Overall survival (OS) | 36 months
  OS, defined as time from first dose of Alkotinib to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Doctor, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China